CLINICAL TRIAL: NCT01222663
Title: Effects of Hemoperfusion With a Polymyxin B Membrane in Peritonitis With Septic Shock
Acronym: ABDO-MIX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meditor SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-67-PMX
Record Dates: First submitted 2010-10-08; First posted 2010-10-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Peritonitis; Septic Shock
Keywords: peritonitis; septic shock; hemoperfusion; Polymyxin B; endotoxin
MeSH Terms: conditions — Peritonitis; Shock, Septic | interventions — Hemoperfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard therapy (Other): Standard therapy in the ICU including but not limited to: antibiotic therapy, nutrition, fluid challenge, vasopressors, hemodynamic monitoring, organ support in the ICU including mechanical ventilation, renal replacement therapy when appropriate
  Interventions: Device: standard therapy
- Hemoperfusion (Experimental): standard therapy + 2 sessions of hemoperfusion within the first 24 hours
  Interventions: Device: standard therapy; Device: hemoperfusion

INTERVENTIONS:
Device: standard therapy — Standard therapy in the ICU including but not limited to: antibiotic therapy, nutrition, fluid challenge, vasopressors, hemodynamic monitoring, organ support in the ICU including mechanical ventilation, renal replacement therapy when appropriate
Device: hemoperfusion — Extracorporeal hemoperfusion with Toraymyxin PMX-20R and conventional medical therapy in the ICU including but not limited to: antibiotic therapy, nutrition, fluid challenge, vasopressors, hemodynamic monitoring, organ support in the ICU including mechanical ventilation, renal replacement therapy when appropriate.
  Other Names: toraymyxin; PMX-20R
  Arms: Hemoperfusion

SUMMARY:
The purpose of this randomized, comparative, open and multi-centre study is to show that two sessions of hemoperfusion with Toraymyxin performed within maximum 36 hours after the surgery of a peritonitis by hollow organ perforation reduce the mortality in patients suffering from septic shock.

DETAILED DESCRIPTION:
The mortality rate due to peritonitis associated to a severe sepsis or a septic shock remains high (between 40 and 60% as per the studies). The recent complementary therapies for severe sepsis have been reassessed (strict glycaemic control, substitutive corticotherapy, activated protein C). Early neutralisation of the endotoxaemia related to gram-negative bacilli sepsis in contact with hemoperfusion membrane covered with polymyxin B (Toraymyxin™) may enable reduction of the inflammatory reaction caused by sepsis and improve its prognosis. 30 studies, including 10 randomized studies, have compared hemoperfusion with Toraymyxin™ to the standard treatment, showing an improvement in the patients' haemodynamic state, oxygenation conditions and reduction in mortality. This treatment is commonly used in Japan. However, the studies conducted either include only a limited number of patients or are not randomized prospective studies. The post-hoc analysis of a recent randomized study conducted on a limited number of patients with abdominal septic shock shows a significant reduction in mortality after factor adjustment. Though the side effects of such a treatment are limited, its cost is high. Hence, extensive prospective studies are necessary to confirm its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed community or nosocomial acquired peritonitis due to organ perforation
* Septic shock requiring catecholamine infusion started or maintained 2 hours after surgery

Exclusion Criteria:

* Pregnancy
* No severity criteria within the 8 hours following surgery
* Neutropenia due to chemotherapy or malignancy
* Abdominal sepsis without peritonitis
* Mesenteric ischemia without perforation
* Peritonitis due to appendicitis
* Perforation linked to trauma
* Cirrhosis child C
* Impossibility to use heparin
* Prolonged cardiac arrest within 72h before surgery
* Terminal disease diagnosed during surgery
* Moribund subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2010-10; Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Mortality | 28 days

SECONDARY OUTCOMES:
organ failure assessed by SOFA score | day 3
delay to withdraw catecholamine after initial shock | day 1-day 28
mortality between the two groups at 7 dayx, 14 days, 21 days and 90 days | 90 days
number of participants with adverse events related to hemoperfusion technique including anticoagulation therapy such as bleeding (type and number of blood transfusion) | day1-day4

CONTACTS AND LOCATIONS:
Overall Officials: Didier Payen, MD, Principal Investigator — Lariboisière University Hospital; René Robert, MD, Principal Investigator — Poitiers University Hospital
Locations (18):
- France (18):
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - Dieppe Hospital, Dieppe
  - Vendée Hospital, La Roche-sur-Yon
  - Dr Schaffner Hospital, Lens
  - Lille University Hospital, Lille
  - Limoges University Hospital, Limoges
  - La Source Hospital, Orléans
  - Lariboisière University Hospital, Paris
  - Saint Louis Hospital, Paris
  - Saint Jean Hospital, Perpignan
  - Bordeaux University Hospital, Pessac
  - Poitiers University Hospital, Poitiers
  - Pontchaillou University Hospital, Rennes
  - Roanne Hospital, Roanne
  - Rouen University Hospital, Rouen
  - Saint-Malo Hospital, St-Malo
  - Strasbourg University Hospital, Strasbourg
  - Tours University Hospital, Tours

REFERENCES:
- [Derived] Payen DM, Guilhot J, Launey Y, Lukaszewicz AC, Kaaki M, Veber B, Pottecher J, Joannes-Boyau O, Martin-Lefevre L, Jabaudon M, Mimoz O, Coudroy R, Ferrandiere M, Kipnis E, Vela C, Chevallier S, Mallat J, Robert R; ABDOMIX Group. Early use of polymyxin B hemoperfusion in patients with septic shock due to peritonitis: a multicenter randomized control trial. Intensive Care Med. 2015 Jun;41(6):975-84. doi: 10.1007/s00134-015-3751-z. Epub 2015 Apr 11. PMID 25862039